CLINICAL TRIAL: NCT07070362
Title: The Construction of a Digital Intelligence Early Warning System for the Whole Process of Acute Lung Injury in Liver Surgery Based on Cardiopulmonary Interaction Characteristics
Brief Title: Digital Early Warning System for Acute Lung Injury in Liver Surgery
Status: Recruiting | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Zhifeng Gao, Chief physician, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: BRWEP2024W032240113; 25254-0-01 (Other: Ethics Committee of Beijing Tsinghua Changgung Hospital)
Record Dates: First submitted 2025-06-11; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Acute Lung Injury(ALI); Liver Cirrhosis; ARDS, Human; MASLD; MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); NAFLD (Nonalcoholic Fatty Liver Disease); Liver Cancer, Adult
Keywords: Digital Intelligence; Acute Lung Injury; PPCs; Liver Surgery; Cardiopulmonary Interaction;
MeSH Terms: conditions — Acute Lung Injury; Liver Cirrhosis; Respiratory Distress Syndrome; Non-alcoholic Fatty Liver Disease; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 3-6ml blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing major liver surgury: Population: 2,497 adult patients (≥18 years) who underwent major liver surgery (≥2 segments resection or transplantation) at Beijing Tsinghua Changgung Hospital, including retrospective (2019.06-2024.05) and prospective (from 2025.12) cohorts.
  Inclusion Criteria: Aged ≥18, scheduled for major liver surgery, with informed consent.
  Exclusion Criteria: Refusal to participate, comorbidities affecting ALI assessment, incomplete data, failed follow-up, or concurrent trials.
  Interventions: None. Observational study; clinical management follows standard protocols without study-related interventions. Data collected from routine records and monitoring.
  Interventions: Other: None-placebo

INTERVENTIONS:
Other: None-placebo — This observational cohort study is non-interventional. Perioperative treatment plans are made based on model - suggested results and anesthesiologists' thought processes, without adding new medicines for patients.

SUMMARY:
This study focuses on developing an explainable machine learning model based on cardiopulmonary interaction characteristics to achieve early prediction of acute lung injury (ALI) in patients undergoing major liver surgery. The research will establish a digital early-warning system for ALI to provide support for clinical diagnosis and treatment decisions, thereby reducing the incidence and fatality rate of ALI.

DETAILED DESCRIPTION:
This study will leverage cardiopulmonary interaction parameters to predict ALI in patients undergoing major liver surgery. Specifically, the research will collect data from preoperative, intraoperative, and postoperative phases. Machine learning algorithms-including logistic regression, random forest, support vector machines (SVM), and neural networks-will be used to develop and validate the prediction model. Model performance will be evaluated using metrics such as accuracy, sensitivity, specificity, and the receiver operating characteristic (ROC) curve. The ultimate objective is to develop a highly accurate and interpretable model that can be integrated into a digital early-warning system for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing major liver surgery (including two-segment or more hepatectomy, liver transplantation, etc.)
* Voluntary participation with signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patient refusal
  * Presence of comorbidities affecting outcome assessment
  * Incomplete outcome records
  * Postoperative follow-up failure
  * Participation in other studies that may interfere with outcome assessment
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of ALI within 7 Days after Surgery | Perioperative period (Perioperative): Refers to the entire process from the determination of surgical treatment to postoperative rehabilitation (e.g., from 1 day before surgery to 7 days after surgery).
  Berlin Definition:
  1. Onset: Acute exacerbation of known injury or new/worsening respiratory symptoms within 1 week.
  2. Chest Imaging (X-ray or CT): Bilateral pulmonary shadows not fully explained by exudation, atelectasis, or nodules.
  3. Pulmonary Edema Etiology: Respiratory failure not fully attributed to heart failure or fluid overload; if no related risk factors, objective tests (e.g., Doppler echocardiography) are needed to exclude hydrostatic pulmonary edema.
  4. Oxygenation Levels: Mild - With CPAP/PEEP >5 cmH2O, 200 mmHg < PaO2/FiO2 < 300 mmHg; Moderate - With CPAP/PEEP >5 cmH2O, 100 mmHg < PaO2/FiO2 < 200 mmHg; Severe - With CPAP/PEEP >5 cmH2O, PaO2/FiO2 < 100 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, School of Clinical Medicine, Tsinghua Medicine，Tsinghua University, Beijing, Beijing Municipality, China

DOCUMENTS (1):
  • Study Protocol (2025-03-27): https://cdn.clinicaltrials.gov/large-docs/62/NCT07070362/Prot_000.pdf